CLINICAL TRIAL: NCT02446327
Title: The Metabolic Road to Diastolic Heart Failure : Diastolic Heart Failure Study (MEDIA-DHF)
Brief Title: The Metabolic Road to Diastolic Heart Failure: Diastolic Heart Failure Study
Acronym: MEDIA-DHF
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Central Hospital, Nancy, France (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2012-A00097-36
Record Dates: First submitted 2015-04-14; First posted 2015-05-18 (Estimated); Last update posted 2015-05-18 (Estimated); Status verified 2015-04

CONDITIONS: Diastolic Heart Failure
MeSH Terms: conditions — Heart Failure, Diastolic | interventions — Blood Specimen Collection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Diastolic heart failure cohort (Other): This is a prospective cohort of patients with diastolic heart failure. Blood sampling for biomarker assessment
  Interventions: Other: Blood sampling for biomarker assessment

INTERVENTIONS:
Other: Blood sampling for biomarker assessment

SUMMARY:
The main objective is to replicate the validation of omics biomarkers of left ventricular diastolic dysfunction in patients with metabolic syndrome.

The aim was to recruit overall 750 patients in Europe (100 for France). Currently, 625 patients were enrolled in Europe and 47 in France.

ELIGIBILITY:
Inclusion Criteria:

* Patients 18 years of age or older
* Signs or symptoms of HF
* Able and willing to provide freely given written informed consent including analysis of genomics

Exclusion Criteria:

* Patients with acute myocardial infarction
* Recent trauma or surgery (< 3 months)
* Hemodynamically significant valvular disease
* Serious cerebrovascular disease or stroke in the last 3 months
* Chronic dialysis
* Chronic liver disease
* Chronic infectious (bacterial or viral) disease
* Any malignant concomitant diseases or a malignant disease in the last 5 years
* Systemic inflammatory diseases, such as autoimmune diseases, connective tissue diseases or collagenoses
* Pregnant women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 47 (Actual)
Dates: Start 2012-01; Primary Completion 2014-03 (Actual); Study Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
Cardiovascular Hospitalizations or Cardiovascular Death | 12 months

SECONDARY OUTCOMES:
Cardiovascular Hospitalizations | 3 months, 6 months, 12 months
Heart Failure Hospitalizations | 3 months, 6 months, 12 months
Other cardiovascular hospitalizations | 3 months, 6 months, 12 months
Non cardiovascular hospitalizations | 3 months, 6 months, 12 months
Cardiovascular Death | 3 months, 6 months, 12 months
Non cardiovascular Death | 3 months, 6 months, 12 months

REFERENCES:
- [Derived] Lagrange J, Jahangiri M PhD, Baudry G, Mercier N, Monzo L, Lamiral Z, Duarte K, Ter Maaten JM, Zannad F, Voors AA, Girerd N. Association Between Endothelial Alterations, Cardiac Function, and Outcomes From Health to Heart Failure: Insight From the STANISLAS, MEDIA-DHF, and BIOSTAT-CHF Cohorts. J Am Heart Assoc. 2025 Jun 3;14(11):e040179. doi: 10.1161/JAHA.124.040179. Epub 2025 May 29. PMID 40439171
- [Derived] Stienen S, Ferreira JP, Kobayashi M, Preud'homme G, Dobre D, Machu JL, Duarte K, Bresso E, Devignes MD, Andres NL, Girerd N, Aakhus S, Ambrosio G, Rocca HB, Fontes-Carvalho R, Fraser AG, van Heerebeek L, de Keulenaer G, Marino P, McDonald K, Mebazaa A, Papp Z, Raddino R, Tschope C, Paulus WJ, Zannad F, Rossignol P. Sex differences in circulating proteins in heart failure with preserved ejection fraction. Biol Sex Differ. 2020 Aug 24;11(1):47. doi: 10.1186/s13293-020-00322-7. PMID 32831121